CLINICAL TRIAL: NCT01278654
Title: Lottery Incentives for Moving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Michael Norton, Associate Professor, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Walkstation2
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Obesity; Sedentary Lifestyle
MeSH Terms: conditions — Obesity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personal incentive (Active Comparator): If participants attain their walkstation usage goal, they are entered into bi-weekly lotteries to win money.
  Interventions: Behavioral: Incentive to exercise
- Token incentive (Active Comparator): Participants who attain their walkstation usage goal will be entered into a bi-weekly prize to win a token reward.
  Interventions: Behavioral: Incentive to exercise

INTERVENTIONS:
Behavioral: Incentive to exercise — Participants who attain their walkstation goal will be entered into a draw every two weeks. We are testing the effect of different prizes on walkstation usage.

SUMMARY:
The purpose of the study is to learn more about effective ways to motivate people to increase their non-exercise energy expenditure exercise. This is an important research question because obesity and weight-related issues are increasingly becoming a problem in America. This project will address this research question by testing the effect of two different incentive schemes in motivating employees who are predominantly sedentary to use Walkstations at work. The Walkstations are treadmills that move at a very slow rate (maximum 2miles / hour) and are attached to a work station (i.e. with computer and telephone); they therefore are designed to increase energy spent not through heavy exercise, but through small changes in posture and movement associated with routines in daily life (called nonexercise activity thermogenesis or NEAT).

Subjects will be employees of Blue Cross Blue Shield of Massachusetts (BCBSMA). Subjects will be the control participants from the previous Walkstation study we ran with BCBSMA. All 120 control participants from this previous study will be told that they can now participate in a study that involves the Walkstations (up until now, they have not been given access to the Walkstations). These participants from the previous study will be sent an email informing them that they are eligible to participate in this new Walkstation pilot. Those who are interested in participating will then be invited to sign up for an enrollment session. There will be no incentives for participating in the initial enrollment session. For the 2 month follow-up session, participants will have a chance to win 1 of 3 prizes (1 * $100, 2 * $50) for completing the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* must pass ParQ

Exclusion Criteria:

* if fail ParQ

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Walkstation usage | after approx 60 days

SECONDARY OUTCOMES:
Biometric measures | baseline and 60 days
  Height, weight, blood pressure
Questionnaire | baseline and 45 days

CONTACTS AND LOCATIONS:
Locations (1):
- Blue Cross Blue Shield Massachusetts, Boston, Massachusetts, United States